CLINICAL TRIAL: NCT04074031
Title: Transcranial Ultrasound Therapy of Essential Tremor
Acronym: ULTRABRAINTher
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190407
Record Dates: First submitted 2019-07-29; First posted 2019-08-29 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-02

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- minimally invasive method for performing thalamotomy (Experimental): We will study patients with essential tremor with significant disability despite well-conducted drug therapy who have a contraindication to deep brain stimulation or who refuse treatment. In this population, unilateral thalamotomy of Vim by radiosurgery is already considered a valid indication and performed routinely with proven efficacy and morbidity deemed acceptable. It is therefore the population of choice to evaluate for the first time in France the efficacy and safety of a new, minimally invasive method for performing thalamotomy: targeted ultrasound thermal injury at high intensity. This same population will also make it possible to study, for the first time in humans in this indication, the potential of neuromodulation by low frequency low frequency ultrasound beams to improve the guidance before the lesion is achieved.
  Interventions: Device: Transcranial Ultrasound Therapy (Exablate® 4000 Type 1.1)

INTERVENTIONS:
Device: Transcranial Ultrasound Therapy (Exablate® 4000 Type 1.1) — The Exablate® 4000 Type 1.1 model designed for noninvasive ablation of brain tissue is an MRI-guided transcranial ultrasound system (MRgFUS). The goal of the Exablate Neuro system is to precisely guide the focus of the ultrasound energy on the target region. The focused ultrasound energy is then repeatedly transmitted to the target until the desired result is achieved. Targeting is performed using MRI acquired during treatment. The treatment process is constantly monitored by closed-loop thermal feedback in real time, under the supervision of the treating physician. Once targeting is complete, the treatment outcome is confirmed by MRI sequences immediately after treatment. The Exablate Neuro is compatible with Siemens 3 Tesla MRI.

SUMMARY:
Context. Essential tremor (ET) is a common disease, disabling in severe forms and resistant to drug treatment. In patients with severe ET, invasive neurosurgical technique such as deep brain stimulation of the Ventral Intermediate (VIM) nucleus of the thalamus is used. Focused ultrasound therapy, creating a small lesion of VIM represents an effective therapeutic alternative of low morbidity with the advantage of not requiring the opening of the skull and penetration into the brain. This therapy is performed under stereotactic guidance. Validation of the target before lesioning is done by testing the clinical effect by a gradual increase in temperature, resulting in tremor reduction. However, the gradual temperature increase in the targeting phase is suboptimal because it can decrease the efficiency of the lesioning procedure. The aim of this research project is to test an innovation of fundamental physics developed by the Langevin Institute, which would allow the reversible modulation of nerve tissue by ultrasonic waves without heating, to predict the effectiveness of treatment of the chosen target within the VIM before creating an irreversible lesion.

Methodology: Fifteen patients with severe and resistant essential tremor will be included in the study. A multimodal MRI will be performed for target calculation using several targeting methods for VIM developed during step 1. For each target, the application of neuro-modulation by ultrasound will allow determine the effect obtained on the tremor (quantified with adequate clinical scales - as Tremor rating scale (CRST), and the recording of electromyographic activity of the upper limbs) and the absence of side effects. A definitive millimetric lesion will be performed at the level of the most relevant target in order to maintain the clinical effect obtained. The procedure will be controlled by thermal MRI sequences. Post-therapy clinical and MRI multimodal follow-up will take place on D1, D7, M1, M2, M3, M6, M12 and M24.

Perspectives and Innovation: This project will test clinically the low intensity ultrasound neuromodulation jointly developed by the Langevin Institute and the Brain and Spine Institute ( ICM) in order to refine the targeting procedure of high intensity transcranial focused ultrasound therapy. In perspective, reversible neuromodulation performed in vivo in humans represents a considerable advance in the exploration and future treatment of neurological and psychiatric diseases such as depression. The translational collaboration between the physicists of the Langevin Institute, the ICM and the medical services of the Pitié-Salpêtrière guarantees the feasibility and quality of this first joint therapeutic trial.

DETAILED DESCRIPTION:
Context:

Essential tremor (ET) is the most common movement disorder, with a prevalence of 1-4% of the general population. ET is characterized by a rapid (6 and 12 Hz) attitude tremor with rhythmic oscillations of agonist and antagonist muscle groups. ET most often affects the upper limbs, the head and the voice but may involve the lower limbs in severe forms. The tremor worsens with age: it extends topographically towards the proximal end of the limbs. In severe forms, drug treatment is ineffective and tremor leads to impaired autonomy.

ET is due to dysfunction of neural networks including the cerebellum, bulbar olive, red nucleus and thalamus nuclei . At the thalamic level, the ventral intermediate thalamic nucleus (VIM), a relay of the cerebellar pathways, is a key structure. This VIM core receives output channels from the cerebellum and projects massively onto the primary motor cortex, the final effector of movement. In humans, imaging studies have shown the involvement of these cerebellar-thalamo-cortical circuits in the pathophysiology of tremor. When drug treatment is ineffective and tremor is disabling, surgical treatments are considered. Deep brain stimulation is the most used reversible and modulable method consisting in implantation of the electrodes in the VIM. However, patients are often elderly with much comorbidity. Thus, in these patients, the act of invasive neurosurgery (neurostimulation) may be contraindicated (anticoagulation treatment) or risky. Also, the peroperative risks such as hematoma of infection exist, even if they are rare.

As an alternative to Deep Brain Stimulation (DBS), radiosurgical thalamotomy was proposed. This method nevertheless has several major disadvantages, such as the use of radioactive sources, the fact that the dose actually delivered during irradiation of the patient cannot be controlled in terms of intensity. On the other hand, the biological effect on the tissues is not immediate and imposes a long waiting time (several months) to evaluate the effectiveness of the treatment. Finally, many cases of radionecrosis have been described with important clinical consequences, although transient in most cases.

Given the limitations inherent to deep brain stimulation and gamma knife thalamotomy, a new method of neuromodulation followed by injury without penetration into the brain would represent a considerable therapeutic hope. In addition, in patients in whom treatment is planned, pre-therapeutic neuromodulation would better determine the target of treatment.

In this context the ultrasonic therapy method was first successfully tested in 2013.These data suggested that the benefit obtained with unilateral ultrasound treatment allows an improvement in tremor comparable to that obtained with deep-brain stimulation of the VIM without significant side effects. More recent series of studies confirmed these initial results with nine studies involving 160 patients in total. These studies have shown a significant clinical improvement with a rate of complication considered as acceptable by the authors (mostly transient ataxia and hemi-chorea-hemiballism) . However, the number of adverse effects remains still rather high and the method of the lesion targeting remains challenging. Also, sometimes it is difficult to obtain the therapeutic effect.

Main objective:

The main objective is the evaluation of the efficacy of transcranial ultrasound treatment, ie the efficacy of the VIM lesion produced by HIFU on contralateral upper extremity tremor in the 3-month procedure.

The secondary objectives are to evaluate:

* the interest of neuromodulation in the change of the initially defined target
* the relevance of the effect of neuromodulation for the prediction of the final clinical effect at 3 and 12 months on controlateral upper extremity tremor at the lesion
* Clinical and accelerometer-mediated symptomatic effects produced by ultrasound neuromodulation of VIM per-procedure
* the safety of ultrasound therapy (HIFU) until one year after the constitution of a unilateral lesion of the intermediate ventral nucleus (VIM) of the thalamus.
* the study of the relationships between precise size and location of the ultrasound-induced lesion and changes in anatomical and functional connectivity and treatment efficacy and side effects.
* the effectiveness of the VIM lesion produced by HIFU on tremor affecting the contralateral upper extremity
* the effectiveness of the VIM lesion produced by HIFU on the overall severity of the tremor
* the effectiveness of HIFU VIM injury on the quality of life of patients with essential tremor
* the overall clinical impression of the patient in terms of severity and evolution compared to the pre-operative state
* the effects of HIFU-induced VIM injury on neurological functions in a global manner
* the effects of HIFU-induced VIM injury on cognitive functions
* the effects of the VIM lesion produced by HIFU on gait and balance
* The study of the structural and functional modifications induced by VIM lesion using structural and functional MRI and its link with therapeutic efficacy.
* neuroanatomical changes and anatomical and functional connectivity The objective of ancillary study: - MRI analysis in diffusion spectroscopy: The investigators team will test the modification of GABAergic and glutamatergic systems of the cerebellum and striatum in TE patients before and after treatment using a newly developed spectroscopic MRI sequence at the neuroimaging center of research of the ICM (CENIR). This new sequence makes it possible to measure the higher-resolution signal in smaller voxels precisely located in the putamen and the cerebellar cortex containing the representation of the limbs. This sequence also makes it possible to obtain a better signal with respect to the noise than the conventional sequences. The investigators team will determine whether the detection of GABA / glutamate abnormalities specific to each region makes it possible to follow the evolution of the patients before and after the ultrasound treatment.

Main steps of work Before the initiation of the ultrasound treatment, the Insightec system will be installed on the Siemens PRISMA MRI at the ICM, CENIR. Adaptation of the Insightec system to the Siemens environment will be performed by the Langevin Institute team, Insightec engineers, and ICM team. The MRI sequences, which are essential for the treatment, will be optimized and adapted to this new environment by concentrating in particular on (i) the correction of the distortions related to the introduction of the probe, and (ii) on the improvement of the spatial resolution. This preliminary work will be done on the phantom and healthy controls for anatomical and temperature sequence optimization.

Fifteen patients with ET will be included in the study. The inclusion and evaluation of patients will take place between 2 months and 2 weeks before the inclusion visit. This visit will verify the inclusion and non-inclusion criteria and provide the information and consent form to the subject. An assessment of the severity of tremor will be made using the CRST scale and electromyographic recordings of the upper limb coupled to functional MRI.

A multimodal MRI scan will be performed for the targeting of the area of interest. Several targeting methods will be performed to have an optimal definition of the target anatomical area. In anatomical sequences, in addition to traditional statistical methods , stereotaxic targeting will be carried out using the three-dimensional and deformable histological atlas of basal ganglia. This atlas allows adapting to the anatomical characteristics of each patient to specifically locate its VIM core. Several methods based on diffusion MRI tractography will also be tested: (i) targeting of the dentato-rubro-thalamic (DRT) pathway connecting the cerebellum to the motor cortex via VIM ; (ii) parcellation of the thalamus using cortical connectivity and (iii) use of the adjacent pathways of the VIM (ML and PT), the VIM being between these pathways. Functional MRI-based methods will also be tested using functional activation MRI to locate the network whose activity is synchronous with tremor electromyographic activity according to a previously developed method.

Patients will be hospitalized in the neurosurgery department for a period of 24 hours. The stereotactic frame will be fixed on the subject's head in the neurosurgery department of the Pitié Salpêtrière under local anesthesia. The CT scan will be performed. Then, the patient will be transferred to CENIR at the ICM. The treatment will take place after placing the focused ultrasound helmet on the MRI bed and installing the subject in the MRI with the helmet.

In the first step, the previously defined targets will be tested using neuro-modulation allowing a transient effect (a few minutes). For each target, the investigators team will determine (i) its level of efficiency through the CRST clinical scale and electromyographic activity of the upper limbs (with electrodes compatible with the MRI environment) and (ii) the absence of side effects (in particular, absence of ipsilateral dystonia, absence of dysarthria, cerebellar ataxia, oculomotor disturbances or sensitivity disorders). In a second step, a final lesion of very small size (1.5x1.5x5mm3) will be performed on the chosen target following the neuro-modulation. The ablation procedure will be controlled by thermal MR sequences.

The visits of the clinical control, including the MRI will take place on D1, D7, M1, M2, M3, M6, M12 and M24. The visits will include general physical examination, collection of current treatments, collection of adverse effects / events, measurement of the severity of tremor: CRST scale, quality of life measurement: Short Form (36) Health Survey : SF-36, assessment of gait and balance: Gait and Balance Scale: GABS, evaluation of cognitive functions, multimodal MRI.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 80
* Diagnosis of essential tremor according to the criteria of the Consensus Statement of the Movement Disorders Society (MDS)
* Patients with significant disability related to their essential Tremor, despite well-conducted medical treatment
* Stable essential tremor drug therapy for at least 30 days prior to inclusion
* Contraindication or refusal or preference of deep brain stimulation
* Patient receiving Social Security or Universal Medical Coverage or any equivalent plan
* Person who voluntarily and knowingly agreed to participate in the study (signing of a written consent)

Exclusion criteria :

* Inability to stop anticoagulant or antiplatelet therapy or any other medication that may increase the risk of bleeding during the 2 weeks prior to the procedure
* Current state of health causing bleeding and / or abnormal coagulopathy
* Unstable cardiac pathology or severe hypertension that cannot be controlled by medication (diastolic blood pressure> 100 with drugs).
* Active epilepsy in the year preceding the inclusion
* Contraindications to magnetic resonance imaging such as non-compatible implanted metal devices (including pacemakers), size limits, etc. including presence of implants in the brain or skull)
* Known hypersensitivity to local anesthetics (Xylocaine 20mg / ml)
* Important claustrophobia that cannot be managed with mild medication
* Inability to maintain prolonged stationary supine position necessary for treatment (3-4 hours)
* Woman of childbearing age without means of contraception
* Pregnant or lactating woman
* Major persons subject to a measure of legal protection (guardianship, curators or under the protection of justice)
* Subject in exclusion period of another biomedical research or participating in any other biomedical stimulation or therapeutic trial
* Patients under AME (state medical aid) (except if exemption from affiliation)
* Patient cannot communicate with the doctor during the treatment procedure
* Subjects with behavior compatible with the abuse of ethanol or psychoactive substances
* Progressive neurological pathology other than TE, stroke or cerebral hemorrhage < 6 months, multiple stroke ATCD, brain tumor or intracranial aneurysm
* Patients who have taken in the last 6 months drugs lowering the epileptogenic threshold significantly (CNS stimulants, sympathomimetics, neuroleptics, imipraminic antidepressants, amantadine, fampridine, fluoroquinolones, mefloquine)
* Significant healing in an area on the path of the planned energy path to the treatment area
* Recourse to neurosurgical treatments for essential tremor (deep brain stimulation or gamma knife

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2024-10-04 (Estimated)

PRIMARY OUTCOMES:
The main objective is to evaluate the efficacy of Vim lesion produced by transcranial focused ultrasound on contralateral upper limb tremor at the 3-month procedure. | 3 MONTHS
  The primary endpoint is the reduction of the severity of essential tremor measured by the clinical assessment of contralateral upper limb tremor at the lesion quantified by CRST A and B at V5 (3 months) compared with V1.

SECONDARY OUTCOMES:
Interest of neuromodulation effect for the prediction of the final clinical effect | 3 MONTHS
  Interest of neuromodulation in the change of the initially defined target in calculating how many times the target has been changed compared to the reference method and therefore the relevance of the neuromodulation effect for the prediction of the final clinical effect at 3 and 12 months on tremor of the upper limb controlateral to the lesion
Adverse events | 24 MONTHS
  The number of adverse events reported or observed between inclusion and the 24th month post-procedure. These events will be collected at all visits from V2 to V8. These events will be classified as sever and non-sever events. They will also be classified as events attributable to the procedure by the medical device, attributable to the lesion or independent of both according to the assumed pathophysiology of the effect.

CONTACTS AND LOCATIONS:
Overall Officials: Nadya Pyatigorskaya, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

REFERENCES:
- [Background] Gallea C, Popa T, Garcia-Lorenzo D, Valabregue R, Legrand AP, Marais L, Degos B, Hubsch C, Fernandez-Vidal S, Bardinet E, Roze E, Lehericy S, Vidailhet M, Meunier S. Intrinsic signature of essential tremor in the cerebello-frontal network. Brain. 2015 Oct;138(Pt 10):2920-33. doi: 10.1093/brain/awv171. Epub 2015 Jun 26. PMID 26115677
- [Background] Bardinet E, Belaid H, Grabli D, Welter ML, Vidal SF, Galanaud D, Derrey S, Dormont D, Cornu P, Yelnik J, Karachi C. Thalamic stimulation for tremor: can target determination be improved? Mov Disord. 2011 Feb 1;26(2):307-12. doi: 10.1002/mds.23448. Epub 2010 Dec 13. PMID 21412838
- [Background] Wintermark M, Druzgal J, Huss DS, Khaled MA, Monteith S, Raghavan P, Huerta T, Schweickert LC, Burkholder B, Loomba JJ, Zadicario E, Qiao Y, Shah B, Snell J, Eames M, Frysinger R, Kassell N, Elias WJ. Imaging findings in MR imaging-guided focused ultrasound treatment for patients with essential tremor. AJNR Am J Neuroradiol. 2014 May;35(5):891-6. doi: 10.3174/ajnr.A3808. Epub 2013 Dec 26. PMID 24371027